CLINICAL TRIAL: NCT05919823
Title: A Phase 3, Multicenter, Two-part Study With a 5-week Double-blind Part (Randomized, Parallel-group, Placebo-controlled) Followed by a 12-week Open-label Extension Part, to Evaluate the Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Chinese Adult Subjects With DSM-5 Schizophrenia
Brief Title: A Study to Assess the Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Chinese Adult Subjects With DSM-5 Schizophrenia
Acronym: UNITE-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CN012-0063; ZL-2701-001 (Other: Zai Lab Protocol ID)
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — Oral xanomeline 50 mg/trospium 20 mg BID on days 1-2 followed by xanomeline 100 mg/trospium 20 mg BID on days 3-7. The dose is increased to xanomeline 125 mg/trospium 30 mg BID on days 8-35 unless the subject is experiencing adverse events from the xanomeline 100 mg/ trospium 20 mg dose. Subjects who were increased to xanomeline 125 mg/trospium 30 mg will have the option to return to xanomeline 100 mg/ trospium 20 mg depending on clinical response and tolerability.
  Other Names: KarXT
  Arms: KarXT
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
A Phase 3, Multicenter, Two-part Study with a 5-week Double-blind Part (Randomized, Parallel-group, Placebo-controlled) followed by a 12-week Open-label Extension Part, to Evaluate the Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Chinese Adult Subjects with DSM-5 Schizophrenia

ELIGIBILITY:
Inclusion Criteria:

1. Subject is Chinese national, aged 18 to 65 years, inclusive, at screening.
2. Subject is capable of providing written informed consent.
3. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 and MINI.
4. Subject is experiencing an acute exacerbation or relapse of psychotic symptoms, with onset less than 2 months before screening.

   1. The subject requires hospitalization for this acute exacerbation or relapse of psychotic symptoms at screen.
   2. If already an inpatient at screening, hospitalization has to be ≤2 weeks for the current exacerbation at the time of screening.
5. PANSS total score between 80 and 120,inclusive, with a scores of ≥4 (moderate or greater) for ≥2 of the following Positive Scale (P) items:

   1. Item 1 (P1; delusions)
   2. Item 2 (P2; conceptual disorganization)
   3. Item 3 (P3; hallucinatory behavior)
   4. Item 6 (P6; suspiciousness/persecution)
6. Subjects with no change (improvement) in PANSS total score between screening and baseline (Day -1) of more than 20%.
7. Subject has a CGI-S score of ≥4 at screening and baseline (Day -1) visits.
8. Subject will have been off lithium therapy for at least 2 weeks before baseline and free of all oral antipsychotic medications for at least 5 half-lives or 1 week, whichever is longer, before baseline (Day -1).
9. Subjects taking a long-acting injectable antipsychotic could not have received a dose of medication for at least 12 weeks (24 weeks for INVEGA TRINZA®) before baseline visit (Day -1).
10. Subject is able to be confined to an inpatient setting for the duration of the 5-week double-blind part of the study, follow instructions, and comply with the protocol requirements.
11. Body mass index of 18 to 40 kg/m2, inclusive.
12. Subject resides in a stable living situation and is anticipated to return to that same stable living situation after discharge, in the opinion of the investigator.
13. Subject has an identified reliable informant. An informant is needed at the screening and baseline visits as well as at the end of the study for relevant assessments (site staff may act as informant while the subject is an inpatient). An informant may not be necessary if the subject has been a patient of the investigator for ≥1 year.
14. Women of childbearing potential (WOCBP) or men whose sexual partners are WOCBP must be willing and able to adhere to the contraception guidelines.

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening).
2. Subjects who are newly diagnosed or are experiencing their first treated episode of schizophrenia.
3. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
4. Subjects with human immunodeficiency virus (HIV), cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on either medical history or liver function test results.
5. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma.
6. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months.
7. Risk for suicidal behavior during the study as determined by the investigator's clinical assessment and C-SSRS.
8. Clinically significant abnormal findings on the physical examination, medical history, electrocardiogram, or clinical laboratory results at screening that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
9. Subjects are receiving or have recently received (within 5 half-lives or 1 week, whichever is longer, before baseline [Day -1]) oral antipsychotic medications; monoamine oxidase inhibitors; anticonvulsants (e.g., lamotrigine, valproate); tricyclic antidepressants (e.g., imipramine, desipramine); selective serotonin reuptake inhibitors; or any other psychoactive medications except for as-needed anxiolytics (e.g., lorazepam, chloral hydrate).
10. Subjects are receiving or have recently received (within 1 week before baseline [Day -1]) metformin.
11. Pregnant, lactating, or less than 3 months postpartum.
12. In the opinion of the investigator and/or Sponsor, subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the investigator and/or Sponsor, may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements.
13. Subject has had psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days before screening.
14. Subject has a history of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) or has required clozapine within the last 12 months.
15. Subjects with prior exposure to KarXT.
16. Subjects who experienced any significant adverse effects due to trospium chloride.
17. Participation in another clinical study within 3 months before screening in which the subject received an experimental or investigational drug agent.
18. Significant risk of violent or destructive behavior.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Anhui Mental Health Center, Hefei, Anhui
  - Wuhu Hospital of Beijing Anding Hospital, Wuhu, Anhui
  - Beijing Anding Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Changping, Beijing Municipality
  - Chongqing 11th People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Mental Health Center, Jiangbei, Chongqing Municipality
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guanzhou, Guangdong
  - The Sixth People's Hosptial of Hebei Province, Baoding, Hebei
  - Daqing City Third Hospital, Daqing, Heilongjiang
  - Zhumadian Second People's Hospital, Zhumadian, Henan
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Jiangxi Mental Health Center, Nanchang, Jiangxi
  - Mental Health Center of Xi'an City, Xi'an, Shaanxi
  - Shandong Mental Health Center, Jinan, Shandong
  - Shandong Daizhuang Hospital, Jining, Shandong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - The Fourth People's Hospital of Chengdu, Chengdu, Sichuan
  - Guangyuan Mental Health Center, Guangyuan, Sichuan
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - Urumqi Fourth People's Hospital, Ürümqi, Xinjiang
  - Hangzhou Seventh People's Hospital, Hangzhou, Zhejiang
  - HuZhou Third Municipal Hospital, Huzhou, Zhejiang
  - Ningbo Kangning Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed 5-week KarXT treatment in the double-blind period and signed ICF for the open-label extension period continued KarXT treatment to additional 12-week.
Groups:
- Double-Blind Part: KarXT: Participants received oral Capsule KarXT (xanomeline 125 mg/trospium 30 mg BID) in a treatment period of 5 weeks. Participants were started on a lead in dose of xanomeline 50 mg/trospium 20 mg twice a day (BID) for the first 2 days followed by xanomeline 100 mg/trospium 20 mg BID for the remainder of Week 1 (Days 3 to 7). On Day 8, dosing was titrated upwards to xanomeline 125 mg/trospium 30 mg BID unless the participant was continuing to experience adverse events from the previous dose increase of xanomeline 100 mg/trospium 20 mg BID. All participants who were increased to xanomeline 125 mg/trospium 30 mg BID, depending on clinical response and tolerability, had the option to return to xanomeline 100 mg/trospium 20 mg BID for the first 3 week of the treatment period.
- Double-Blind Part: Placebo: Participants received the matching placebo to KarXT orally twice daily for a treatment period of 5 weeks.
- Open-Label Part: KarXT/KarXT: Participants completed 5-week KarXT treatment in the double-blind part and signed ICF for the open-label part. Participants continued oral Capsule KarXT (xanomeline 125 mg/trospium 30 mg BID) in a long-term treatment period of 12 weeks. In the open-label part, participants were started on a lead in dose of xanomeline 50 mg/trospium 20 mg twice a day (BID) for the first 2 days followed by xanomeline 100 mg/trospium 20 mg BID for the remainder of Week (Days 3 to 7) of the open-label part. On Day 8, dosing was titrated upwards to xanomeline 125 mg/trospium 30 mg BID unless the participant was continuing to experience adverse events from the previous dose increase of xanomeline 100 mg/trospium 20 mg BID. All participants who were increased to xanomeline 125 mg/trospium 30 mg BID, depending on clinical response and tolerability, had the option to return to xanomeline 100 mg/trospium 20 mg BID for the remainder of the treatment period.
- Open-Label Part: Placebo/KarXT: Participants completed 5-week matching placebo to KarXT in the double-blind part and signed ICF for the open-label part. Participants continued oral Capsule KarXT (xanomeline 125 mg/trospium 30 mg BID) in a long-term treatment period of 12 weeks. In the open-label part, participants were started on a lead in dose of xanomeline 50 mg/trospium 20 mg twice a day (BID) for the first 2 days followed by xanomeline 100 mg/trospium 20 mg BID for the remainder of Week (Days 3 to 7) of the open-label part. On Day 8, dosing was titrated upwards to xanomeline 125 mg/trospium 30 mg BID unless the participant was continuing to experience adverse events from the previous dose increase of xanomeline 100 mg/trospium 20 mg BID. All participants who were increased to xanomeline 125 mg/trospium 30 mg BID, depending on clinical response and tolerability, had the option to return to xanomeline 100 mg/trospium 20 mg BID for the remainder of the treatment period.
Period: Pre-Treatment Period
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Started (Started = randomized) | 103 | 99 | 0 | 0
Completed (Completed = treated) | 102 | 98 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Double-Blind Period
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Started (Started = Started the 5-week double-blind period) | 102 | 98 | 0 | 0
Completed (Completed = Completed the 5-week double-blind period) | 79 | 78 | 0 | 0
Not Completed | 23 | 20 | 0 | 0
Not completed — Adverse Event | 8 | 9 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Participant withdrew consent | 11 | 7 | 0 | 0
Not completed — Other reasons | 2 | 3 | 0 | 0
Period: Open Label Period
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Started (Started = Completed double-blind period and Started 12-week open label period.) | 0 | 0 | 38 (Not all participants who completed the double-blind period started in the open-label period.) | 28 (Not all participants who completed the double-blind period started in the open-label period.)
Completed (Completed = Completed 12 week-open label period.) | 0 | 0 | 18 | 11
Not Completed | 0 | 0 | 20 | 17
Not completed — Adverse Event | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Participant withdrew consent | 0 | 0 | 8 | 6
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Other reasons | 0 | 0 | 9 | 5

BASELINE CHARACTERISTICS:
Population: Open-Label participants are accounted for under their Double-Blind Groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT | Total
Number analyzed (Participants) | 103 | 99 | 0 | 0 | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (9.55) | 36.9 (11.91) |  |  | 37.1 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 50 |  |  | 106
  Male | 47 | 49 |  |  | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  |  | 0
  Not Hispanic or Latino | 103 | 99 |  |  | 202
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 103 | 99 |  |  | 202
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 0 | 0 |  |  | 0
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Scores at Week 5 of the Double-Blind Period
Description: PANSS Total Score is a clinical tool used to measure the severity of symptoms in individuals with schizophrenia. It includes 30 items divided into three subscales:
  Positive Symptoms (e.g., hallucinations, delusions) Negative Symptoms (e.g., social withdrawal, lack of motivation) General Psychopathology (e.g., anxiety, depression) Each item is rated from 1 (absent) to 7 (extreme), resulting in a total score range from 30 to 210.
  Higher PANSS Total Scores indicate more severe symptoms and worse clinical outcomes.
  Baseline is defined as last non-missing assessment prior to the first dose of study drug.
Time Frame: At Baseline and at Week 5 of the Double-Blind Period
Population: All randomized participants who received at least one dose of study medicine and had baseline and least 1 post-baseline PANSS assessment in the double-blind period. Prespecified to be reported for the double-blind period only.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 99 | 97
Score on a Scale | -16.9 (2.122) | -7.7 (2.074)
Statistical Analysis 1: Comparison: Double-Blind Part: KarXT vs Double-Blind Part: Placebo; Test type: Superiority — Least-squares mean difference; p = 0.0014, Mixed model repeated measure; MMRM includes PANSS change at Weeks 2-5; fixed effects: treatment, visit, interaction; covariates: site, age, sex, baseline; Least-squares mean difference = -9.2, 95% CI 2-sided [-14.8 to -3.6], Standard Error of Mean 2.835 — Numerator=KarXT/KarXT, denominator =Placebo/KarXT

2. Secondary Outcome: Change From Baseline in Positive Symptom Score of the Positive and Negative Syndrome Scale (PANSS) at Week 5 of the Double-Blind Period
Description: The PANSS Positive Symptom Score assesses the severity of positive symptoms in schizophrenia, such as hallucinations and delusions. It includes 7 items: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. Each item is rated from 1 (absent) to 7 (extreme), for a total score range of 7 to 49. Higher scores indicate more severe symptoms and worse clinical outcomes.
  Baseline is defined as last non-missing assessment prior to the first dose of study drug.
Time Frame: At Baseline and at Week 5 of the Double-Blind Period
Population: All randomized participants who received at least one dose of study medicine and had baseline and least 1 post-baseline PANSS assessment in the double-blind period. Prespecified to be collected for the double-blind period only.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 99 | 97
Score on a Scale | -6.5 (0.713) | -4.6 (0.700)
Statistical Analysis 1: Comparison: Double-Blind Part: KarXT vs Double-Blind Part: Placebo; Test type: Superiority — Least-squares mean difference; p = 0.0474, Mixed model for Repeated measures; includes PANSS change at Weeks 2-5; fixed effects: treatment, visit, interaction; covariates: site, age, sex, baseline PANSS positive symptom score; Least-squares mean difference = -1.9, 95% CI 2-sided [-3.8 to 0], Standard Error of Mean 0.952 — Numerator=KarXT/KarXT, denominator =Placebo/KarXT

3. Secondary Outcome: Change From Baseline in Negative Symptom Score of the Positive and Negative Syndrome Scale (PANSS) at Week 5 of the Double-Blind Period
Description: The Positive and Negative Syndrome Scale (PANSS) Negative Symptom Score assesses the severity of negative symptoms in schizophrenia, such as emotional withdrawal and reduced motivation. It includes 7 items: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity, and stereotyped thinking. Each item is rated from 1 (absent) to 7 (extreme), for a total score range of 7 to 49. Higher scores indicate more severe symptoms and worse outcomes.
  Baseline is defined as last non-missing assessment prior to the first dose of study drug.
Time Frame: At Baseline and at Week 5 of the Double-Blind Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 99 | 97
Score on a Scale | -3.2 (0.664) | -0.7 (0.648)
Statistical Analysis 1: Comparison: Double-Blind Part: KarXT vs Double-Blind Part: Placebo; Test type: Superiority — Least-squares mean difference; p = 0.0062, Mixed model for Repeated measures; [statistical method as in outcome 2, analysis 1]; Least-squares mean difference = -2.5, 95% CI 2-sided [-4.2 to -0.7], Standard Error of Mean 0.887

4. Secondary Outcome: Change From Baseline in Negative Marder Factor Score of the Positive and Negative Syndrome Scale (PANSS) at Week 5 of the Double-Blind Period
Description: The Negative Marder Factor Score is subset of PANSS items used to evaluate negative symptoms based on a five-factor model. It includes 7 items: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of spontaneity, motor retardation, and active social avoidance. Each item is rated from 1 to 7. Higher scores reflect greater severity of negative symptoms and poorer clinical outcomes. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms. The PANSS Total Score is then the sum of the positive, negative, and general psychopathology symptom scores. Baseline is defined as last non-missing assessment prior to the first dose of study drug.
Time Frame: At Baseline and at Week 5 of the Double-Blind Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 99 | 97
Score on a Scale | -3.1 (0.677) | -0.5 (0.660)
Statistical Analysis 1: Comparison: Double-Blind Part: KarXT vs Double-Blind Part: Placebo; Test type: Superiority — Least-squares mean difference; p = 0.0056, Mixed model for Repeated measures; [statistical method as in outcome 2, analysis 1]; Least-squares mean difference = -2.5, 95% CI 2-sided [-4.3 to -0.8], Standard Error of Mean 0.906

5. Secondary Outcome: Change From Baseline in Clinical Global Impressions - Severity (CGI-S) Score at Week 5 of the Double-Blind Period
Description: The CGI-S Score is a clinician-rated scale used to assess the severity of a patient's mental illness at a given time. It ranges from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients). The score reflects the clinician's overall impression based on observed symptoms, behavior, and functioning. Higher scores indicate greater illness severity and worse clinical status.
  Baseline is defined as last non-missing assessment prior to the first dose of study drug.
Time Frame: At Baseline and at Week 5 of the Double-Blind Period
Population: All randomized participants who received at least one dose of study medicine and had baseline and least 1 post-baseline CGI-S assessment in the double-blind period. Prespecified to be reported for the double-blind period only.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 99 | 97
Score on a Scale | -0.9 (0.119) | -0.5 (0.117)
Statistical Analysis 1: Comparison: Double-Blind Part: KarXT vs Double-Blind Part: Placebo; Test type: Superiority — Least-squares mean difference; p = 0.0208, Mixed model for repeated measures; ncludes PANSS change at Weeks 2-5; fixed effects: treatment, visit, interaction; covariates: site, age, sex, baseline PANSS positive symptom score; Least-squares mean difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.165

6. Secondary Outcome: Percentage of PANSS Responders (≥30% Change in PANSS Total Score From Baseline) at Week 5 of the Double-Blind Period
Description: as for outcome 1
Time Frame: At Baseline and at Week 5 of the Double-Blind Period
Population: All randomized participants who received at least one dose of study medicine and had baseline and least 1 post-baseline PANSS assessment (≥30% Change) in the double-blind period. Prespecified to be reported for the double-blind period only.
Measure: Number; unit: Percentage of participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 76 | 76
Percentage of participants | 42.1 | 26.3
Statistical Analysis 1: Comparison: Double-Blind Part: KarXT vs Double-Blind Part: Placebo; Test type: Superiority; p = 0.0402, Chi-squared; Percentage difference = 15.8, 95% CI 2-sided [0.7 to 29.9]

7. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Scores at Week 12 of the Open-Label Period
Description: PANSS Total Score is a clinical tool used to measure the severity of symptoms in individuals with schizophrenia. It includes 30 items divided into three subscales:
  Positive Symptoms (e.g., hallucinations, delusions) Negative Symptoms (e.g., social withdrawal, lack of motivation) General Psychopathology (e.g., anxiety, depression) Each item is rated from 1 (absent) to 7 (extreme), resulting in a total score range from 30 to 210.
  Higher PANSS Total Scores indicate more severe symptoms and worse clinical outcomes.
  Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At Baseline and at Week 12 of the Open-Label Period
Population: All participants who received at least one dose of study medicine in the open-label period and had study/open-label period baseline and least 1 post-baseline PANSS assessment in the Open-label Period. Prespecified to be reported for the open-label period only.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 18 | 11
Score on a Scale
  Study baseline to Open-label period- Week 12 | -22.0 (21.67) | -21.2 (19.76)
  Open-label period- baseline to Open-label period- Week 12 | -2.7 (17.27) | -6.1 (12.49)

8. Secondary Outcome: Change From Baseline in Positive Symptom Score of the Positive and Negative Syndrome Scale (PANSS) at Week 12 of the Open-Label Period
Description: The PANSS Positive Symptom Score assesses the severity of positive symptoms in schizophrenia, such as hallucinations and delusions. It includes 7 items: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. Each item is rated from 1 (absent) to 7 (extreme), for a total score range of 7 to 49. Higher scores indicate more severe symptoms and worse clinical outcomes.
  Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At Baseline and at Week 12 of the Open-Label Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 18 | 11
Score on a Scale
  Study baseline to Open-label period - Week 12 | -6.9 (6.09) | -8.2 (6.65)
  Open-label period- baseline to Open-label period- Week 12 | -0.2 (5.31) | -0.8 (4.64)

9. Secondary Outcome: Change From Baseline in Negative Symptom Score of the Positive and Negative Syndrome Scale (PANSS) at Week 12 of the Open-Label Period
Description: The Positive and Negative Syndrome Scale (PANSS) Negative Symptom Score assesses the severity of negative symptoms in schizophrenia, such as emotional withdrawal and reduced motivation. It includes 7 items: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity, and stereotyped thinking. Each item is rated from 1 (absent) to 7 (extreme), for a total score range of 7 to 49. Higher scores indicate more severe symptoms and worse outcomes.
  Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At Baseline and at Week 12 of the Open-Label Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 18 | 11
Score on a Scale
  Study baseline to Open-label period- Week 12 | -4.3 (7.75) | -3.0 (7.40)
  Open-label period- baseline to Open-label period- Week 12 | -0.4 (5.64) | -1.4 (4.88)

10. Secondary Outcome: Change From Baseline in Negative Marder Factor Score of the Positive and Negative Syndrome Scale (PANSS) at Week 12 of the Open-Label Period
Description: The Negative Marder Factor Score is subset of PANSS items used to evaluate negative symptoms based on a five-factor model. It includes 7 items: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of spontaneity, motor retardation, and active social avoidance. Each item is rated from 1 to 7. Higher scores reflect greater severity of negative symptoms and poorer clinical outcomes.
  Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At Baseline and at Week 12 of the Open-Label Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 18 | 11
Score on a Scale
  Study baseline to Open-label period- Week 12 | -3.9 (7.40) | -3.0 (7.25)
  Open-label period- baseline to Open-label period- Week 12 | -0.2 (5.43) | -0.8 (4.49)

11. Secondary Outcome: Change From Baseline in Clinical Global Impressions - Severity (CGI-S) Score at Week 12 of the Open-Label Period
Description: The CGI-S Score is a clinician-rated scale used to assess the severity of a patient's mental illness at a given time. It ranges from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients). The score reflects the clinician's overall impression based on observed symptoms, behavior, and functioning. Higher scores indicate greater illness severity and worse clinical status.
  Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At Baseline and at Week 12 of the Open-Label Period
Population: All participants who received at least one dose of study medicine in the open-label period and had study/open-label period baseline and least 1 post-baseline CGI-S assessment in the Open-label Period. Prespecified to be reported for the open-label period only.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 18 | 11
Score on a Scale
  Study baseline to Open-label period- Week 12 | -1.1 (1.06) | -1.2 (0.98)
  Open-label period- baseline to Open-label period- Week 12 | -0.1 (0.80) | -0.5 (0.82)

12. Secondary Outcome: Percentage of PANSS Responders (≥30% Change in PANSS Total Score From Baseline) at Week 12 of the Open-Label Period
Description: as for outcome 7
Time Frame: At Baseline and at Week 12 of the Open-Label Period
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 18 | 11
Percentage of participants
  Study baseline to Open-label period- Week 12 | 66.7 | 45.5
  Open-label period- baseline to Open-label period- Week 12 | 16.7 | 27.3

13. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Study Drug Withdrawal
Description: Adverse Event (AE):
  An AE is any unfavorable and unintended sign, symptom, or disease that occurs in a participant during a clinical trial, regardless of whether it is related to the study treatment. This includes new conditions or worsening of pre-existing ones.
  Serious Adverse Event (SAE):
  An SAE is an AE that results in death, is life-threatening, requires hospitalization or prolongs existing hospitalization, causes persistent or significant disability/incapacity, or leads to a congenital anomaly/birth defect. Other events may be considered serious if they require medical intervention to prevent one of these outcomes.
Time Frame: From first dose until study completion (up to approximately 18 weeks)
Population: All treated participants in the double blind/open-label periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 102 | 98 | 38 | 28
Participants
  Adverse events | 97 | 90 | 33 | 28
  Serious adverse events | 0 | 3 | 0 | 3
  Adverse events leading to drug withdrawal | 8 | 9 | 2 | 4

14. Secondary Outcome: Number of Participants With Orthostatic Vital Sign Events
Description: Orthostatic vital signs included blood pressure and heart rate. A participant having sustained orthostatic event is defined as the participant experienced at least one orthostatic event for at least 3 consecutive visits.
Time Frame: From first dose until study completion (up to approximately 18 weeks)
Population: All treated participants in the double blind/open-label periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 102 | 98 | 38 | 28
Participants
  Orthostatic event at any visit | 36 | 31 | 8 | 5
  A Decrease in Systolic Blood Pressure of ≥ 20 mmHg | 21 | 10 | 2 | 2
  A Decrease in Diastolic Blood Pressure of ≥ 10 mmHg | 16 | 16 | 4 | 5
  An Increase in Heart Rate of ≥ 30 bpm | 9 | 12 | 2 | 0
  Sustained orthostatic events | 3 | 2 | 0 | 0

15. Secondary Outcome: Number of Participants With Elevated Liver Function Test Results
Description: ULN = upper limit of normal range.; DB = Double-blind period; OL = Open-label period. Hy's law is defined as an elevated alanine aminotransferase level (>3xULN) or an elevated aspartate aminotransferase (>3xULN) in combination with alkaline phosphatase <2xULN and elevated total bilirubin (>2 x ULN). Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At study baseline, Day 21 DB, Day 35 DB, open-label baseline, Day 14 OL, Day 84 OL, and end of study visit (up to approximately 18 weeks)
Population: All treated participants with baseline and at least one post baseline liver function assessment in the double blind/open-label periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 102 | 98 | 38 | 28
Participants
  Study Baseline - Alanine aminotransferase - >3XULN | 0 | 0 | 0 | 0
  Study Baseline - Alanine aminotransferase - >5XULN | 0 | 0 | 0 | 0
  Study Baseline - Alanine aminotransferase - >8XULN | 0 | 0 | 0 | 0
  Study Baseline - Alanine aminotransferase - >10XULN | 0 | 0 | 0 | 0
  Study Baseline - Alanine aminotransferase - >20XULN | 0 | 0 | 0 | 0
  Study Baseline - Aspartate Aminotransferase - >3XULN | 0 | 0 | 0 | 0
  Study Baseline - Aspartate Aminotransferase - >5XULN | 0 | 0 | 0 | 0
  Study Baseline - Aspartate Aminotransferase - >8XULN | 0 | 0 | 0 | 0
  Study Baseline - Aspartate Aminotransferase - >10XULN | 0 | 0 | 0 | 0
  Study Baseline - Aspartate Aminotransferase - >20XULN | 0 | 0 | 0 | 0
  Study Baseline - Alkaline phosphatase - >1.5XULN | 0 | 0 | 0 | 0
  Study Baseline - Alkaline phosphatase - >2XULN | 0 | 0 | 0 | 0
  Study Baseline - Bilirubin - >1.5XULN | 0 | 2 | 0 | 1
  Study Baseline - Bilirubin - >2XULN | 0 | 0 | 0 | 0
  Study Baseline - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 101 | 98 | 38 | 28
  Study Baseline - Gamma glutamyl transferase - >2XULN | 1 | 1 | 1 | 0
  Study Baseline - Hy's law cases | 0 | 0 | 0 | 0
  Day 21 DB - Alanine aminotransferase - >3XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alanine aminotransferase - >3XULN | 5 | 0 |  |
  Day 21 DB - Alanine aminotransferase - >5XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alanine aminotransferase - >5XULN | 2 | 0 |  |
  Day 21 DB - Alanine aminotransferase - >8XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alanine aminotransferase - >8XULN | 1 | 0 |  |
  Day 21 DB - Alanine aminotransferase - >10XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alanine aminotransferase - >10XULN | 0 | 0 |  |
  Day 21 DB - Alanine aminotransferase - >20XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alanine aminotransferase - >20XULN | 0 | 0 |  |
  Day 21 DB - Aspartate Aminotransferase - >3XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Aspartate Aminotransferase - >3XULN | 1 | 0 |  |
  Day 21 DB - Aspartate Aminotransferase - >5XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Aspartate Aminotransferase - >5XULN | 1 | 0 |  |
  Day 21 DB- Aspartate Aminotransferase - >8XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB- Aspartate Aminotransferase - >8XULN | 1 | 0 |  |
  Day 21 DB - Aspartate Aminotransferase - >10XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Aspartate Aminotransferase - >10XULN | 1 | 0 |  |
  Day 21 DB - Aspartate Aminotransferase - >20XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Aspartate Aminotransferase - >20XULN | 0 | 0 |  |
  Day 21 DB - Alkaline phosphatase - >1.5XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alkaline phosphatase - >1.5XULN | 2 | 0 |  |
  Day 21 DB - Alkaline phosphatase - >2XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Alkaline phosphatase - >2XULN | 0 | 0 |  |
  Day 21 DB - Bilirubin - >1.5XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Bilirubin - >1.5XULN | 0 | 2 |  |
  Day 21 DB - Bilirubin - >2XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Bilirubin - >2XULN | 0 | 0 |  |
  Day 21 DB - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Gamma glutamyl transferase - >2XULN | 9 | 1 |  |
  Day 21 DB - Hy's law cases: number analyzed (Participants) | 88 | 91 | 0 | 0
  Day 21 DB - Hy's law cases | 0 | 0 |  |
  Day 35 DB - Alanine aminotransferase - >3XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alanine aminotransferase - >3XULN | 0 | 1 |  |
  Day 35 DB - Alanine aminotransferase - >5XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alanine aminotransferase - >5XULN | 0 | 0 |  |
  Day 35 DB - Alanine aminotransferase - >8XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alanine aminotransferase - >8XULN | 0 | 0 |  |
  Day 35 DB - Alanine aminotransferase - >10XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alanine aminotransferase - >10XULN | 0 | 0 |  |
  Day 35 DB - Alanine aminotransferase - >20XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alanine aminotransferase - >20XULN | 0 | 0 |  |
  Day 35 DB - Aspartate Aminotransferase - >3XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Aspartate Aminotransferase - >3XULN | 0 | 0 |  |
  Day 35 DB - Aspartate Aminotransferase - >5XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Aspartate Aminotransferase - >5XULN | 0 | 0 |  |
  Day 35 DB - Aspartate Aminotransferase - >8XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Aspartate Aminotransferase - >8XULN | 0 | 0 |  |
  Day 35 DB - Aspartate Aminotransferase - >10XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Aspartate Aminotransferase - >10XULN | 0 | 0 |  |
  Day 35 DB - Aspartate Aminotransferase - >20XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Aspartate Aminotransferase - >20XULN | 0 | 0 |  |
  Day 35 DB - Alkaline phosphatase - >1.5XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alkaline phosphatase - >1.5XULN | 0 | 1 |  |
  Day 35 DB - Alkaline phosphatase - >2XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Alkaline phosphatase - >2XULN | 0 | 1 |  |
  Day 35 DB - Bilirubin - >1.5XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Bilirubin - >1.5XULN | 0 | 4 |  |
  Day 35 DB - Bilirubin - >2XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Bilirubin - >2XULN | 0 | 0 |  |
  Day 35 DB - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Gamma glutamyl transferase - >2XULN | 3 | 2 |  |
  Day 35 DB - Hy's law cases: number analyzed (Participants) | 80 | 78 | 0 | 0
  Day 35 DB - Hy's law cases | 0 | 0 |  |
  End of study - Alanine aminotransferase - >3XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alanine aminotransferase - >3XULN | 0 | 0 | 0 | 0
  End of study - Alanine aminotransferase - >5XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alanine aminotransferase - >5XULN | 0 | 0 | 0 | 0
  End of study - Alanine aminotransferase - >8XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alanine aminotransferase - >8XULN | 0 | 0 | 0 | 0
  End of study - Alanine aminotransferase - >10XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alanine aminotransferase - >10XULN | 0 | 0 | 0 | 0
  End of study - Alanine aminotransferase - >20XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alanine aminotransferase - >20XULN | 0 | 0 | 0 | 0
  End of study - Aspartate Aminotransferase - >3XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Aspartate Aminotransferase - >3XULN | 0 | 0 | 0 | 0
  End of study - Aspartate Aminotransferase - >5XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Aspartate Aminotransferase - >5XULN | 0 | 0 | 0 | 0
  End of study - Aspartate Aminotransferase - >8XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Aspartate Aminotransferase - >8XULN | 0 | 0 | 0 | 0
  End of study - Aspartate Aminotransferase - >10XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Aspartate Aminotransferase - >10XULN | 0 | 0 | 0 | 0
  End of study - Aspartate Aminotransferase - >20XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Aspartate Aminotransferase - >20XULN | 0 | 0 | 0 | 0
  End of study - Alkaline phosphatase - >1.5XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alkaline phosphatase - >1.5XULN | 0 | 1 | 0 | 0
  End of study - Alkaline phosphatase - >2XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Alkaline phosphatase - >2XULN | 0 | 0 | 0 | 0
  End of study - Bilirubin - >1.5XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Bilirubin - >1.5XULN | 0 | 0 | 0 | 0
  End of study - Bilirubin - >2XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Bilirubin - >2XULN | 0 | 0 | 0 | 0
  End of study - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Gamma glutamyl transferase - >2XULN | 1 | 1 | 0 | 0
  End of study - Hy's law cases: number analyzed (Participants) | 43 | 40 | 38 | 28
  End of study - Hy's law cases | 0 | 0 | 0 | 0
  Open-label baseline - Alanine aminotransferase - >3XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alanine aminotransferase - >3XULN |  |  | 0 | 0
  Open-label baseline - Alanine aminotransferase - >5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alanine aminotransferase - >5XULN |  |  | 0 | 0
  Open-label baseline - Alanine aminotransferase - >8XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alanine aminotransferase - >8XULN |  |  | 0 | 0
  Open-label baseline - Alanine aminotransferase - >10XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alanine aminotransferase - >10XULN |  |  | 0 | 0
  Open-label baseline - Alanine aminotransferase - >20XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alanine aminotransferase - >20XULN |  |  | 0 | 0
  Open-label baseline - Aspartate Aminotransferase - >3XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Aspartate Aminotransferase - >3XULN |  |  | 0 | 0
  Open-label baseline - Aspartate Aminotransferase - >5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Aspartate Aminotransferase - >5XULN |  |  | 0 | 0
  Open-label baseline - Aspartate Aminotransferase - >8XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Aspartate Aminotransferase - >8XULN |  |  | 0 | 0
  Open-label baseline - Aspartate Aminotransferase - >10XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Aspartate Aminotransferase - >10XULN |  |  | 0 | 0
  Open-label baseline - Aspartate Aminotransferase - >20XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Aspartate Aminotransferase - >20XULN |  |  | 0 | 0
  Open-label baseline - Alkaline phosphatase - >1.5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alkaline phosphatase - >1.5XULN |  |  | 0 | 0
  Open-label baseline - Alkaline phosphatase - >2XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Alkaline phosphatase - >2XULN |  |  | 0 | 0
  Open-label baseline - Bilirubin - >1.5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Bilirubin - >1.5XULN |  |  | 0 | 0
  Open-label baseline - Bilirubin - >2XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Bilirubin - >2XULN |  |  | 0 | 0
  Open-label baseline - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Gamma glutamyl transferase - >2XULN |  |  | 1 | 0
  Open-label baseline - Hy's law cases: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Hy's law cases |  |  | 0 | 0
  Day 14 OL - Alanine aminotransferase - >3XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alanine aminotransferase - >3XULN |  |  | 1 | 0
  Day 14 OL - Alanine aminotransferase - >5XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alanine aminotransferase - >5XULN |  |  | 0 | 0
  Day 14 OL - Alanine aminotransferase - >8XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alanine aminotransferase - >8XULN |  |  | 0 | 0
  Day 14 OL - Alanine aminotransferase - >10XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alanine aminotransferase - >10XULN |  |  | 0 | 0
  Day 14 OL - Alanine aminotransferase - >20XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alanine aminotransferase - >20XULN |  |  | 0 | 0
  Day 14 OL - Aspartate Aminotransferase - >3XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Aspartate Aminotransferase - >3XULN |  |  | 0 | 0
  Day 14 OL - Aspartate Aminotransferase - >5XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Aspartate Aminotransferase - >5XULN |  |  | 0 | 0
  Day 14 OL - Aspartate Aminotransferase - >8XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Aspartate Aminotransferase - >8XULN |  |  | 0 | 0
  Day 14 OL - Aspartate Aminotransferase - >10XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Aspartate Aminotransferase - >10XULN |  |  | 0 | 0
  Day 14 OL - Aspartate Aminotransferase - >20XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Aspartate Aminotransferase - >20XULN |  |  | 0 | 0
  Day 14 OL - Alkaline phosphatase - >1.5XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alkaline phosphatase - >1.5XULN |  |  | 0 | 0
  Day 14 OL - Alkaline phosphatase - >2XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Alkaline phosphatase - >2XULN |  |  | 0 | 0
  Day 14 OL - Bilirubin - >1.5XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Bilirubin - >1.5XULN |  |  | 0 | 0
  Day 14 OL - Bilirubin - >2XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Bilirubin - >2XULN |  |  | 0 | 0
  Day 14 OL - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Gamma glutamyl transferase - >2XULN |  |  | 1 | 0
  Day 14 OL - Hy's law cases: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Hy's law cases |  |  | 0 | 0
  Day 84 - OL - Alanine aminotransferase - >3XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alanine aminotransferase - >3XULN |  |  | 0 | 0
  Day 84 - OL - Alanine aminotransferase - >5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alanine aminotransferase - >5XULN |  |  | 0 | 0
  Day 84 - OL - Alanine aminotransferase - >8XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alanine aminotransferase - >8XULN |  |  | 0 | 0
  Day 84 - OL - Alanine aminotransferase - >10XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alanine aminotransferase - >10XULN |  |  | 0 | 0
  Day 84 - OL - Alanine aminotransferase - >20XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alanine aminotransferase - >20XULN |  |  | 0 | 0
  Day 84 - OL - Aspartate Aminotransferase - >3XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Aspartate Aminotransferase - >3XULN |  |  | 0 | 0
  Day 84 - OL - Aspartate Aminotransferase - >5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Aspartate Aminotransferase - >5XULN |  |  | 0 | 0
  Day 84 - OL - Aspartate Aminotransferase - >8XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Aspartate Aminotransferase - >8XULN |  |  | 0 | 0
  Day 84 - OL - Aspartate Aminotransferase - >10XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Aspartate Aminotransferase - >10XULN |  |  | 0 | 0
  Day 84 - OL - Aspartate Aminotransferase - >20XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Aspartate Aminotransferase - >20XULN |  |  | 0 | 0
  Day 84 - OL - Alkaline phosphatase - >1.5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alkaline phosphatase - >1.5XULN |  |  | 0 | 0
  Day 84 - OL - Alkaline phosphatase - >2XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Alkaline phosphatase - >2XULN |  |  | 0 | 0
  Day 84 - OL - Bilirubin - >1.5XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Bilirubin - >1.5XULN |  |  | 0 | 0
  Day 84 - OL - Bilirubin - >2XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Bilirubin - >2XULN |  |  | 0 | 0
  Day 84 - OL - Gamma glutamyl transferase - >2XULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Gamma glutamyl transferase - >2XULN |  |  | 0 | 0
  Day 84 - OL - Hy's law cases: number analyzed (Participants) | 0 | 0 | 38 | 28
  Day 84 - OL - Hy's law cases |  |  | 0 | 0

16. Secondary Outcome: Number of Participants With Elevated Metabolic Syndrome Parameters
Description: ULN = Upper limit of normal; DB = Double-blind period; OL = Open-label period. Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: as for outcome 15
Population: All treated participants with baseline and at least one post-baseline result in the double blind/open-label periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 102 | 98 | 38 | 28
Participants
  Study baseline - Glucose > ULN | 14 | 18 | 6 | 8
  Study baseline - Total Cholesterol > ULN | 19 | 11 | 6 | 5
  Study baseline - Triglycerides > ULN | 18 | 20 | 5 | 8
  Day 21 DB - Glucose > ULN: number analyzed (Participants) | 88 | 90 | 0 | 0
  Day 21 DB - Glucose > ULN | 10 | 8 |  |
  Day 21 DB - Total Cholesterol > ULN: number analyzed (Participants) | 88 | 90 | 0 | 0
  Day 21 DB - Total Cholesterol > ULN | 7 | 6 |  |
  Day 21 DB - Triglycerides > ULN: number analyzed (Participants) | 88 | 90 | 0 | 0
  Day 21 DB - Triglycerides > ULN | 19 | 22 |  |
  Day 35 DB - Glucose > ULN: number analyzed (Participants) | 81 | 78 | 0 | 0
  Day 35 DB - Glucose > ULN | 12 | 12 |  |
  Day 35 DB - Total Cholesterol > ULN: number analyzed (Participants) | 81 | 78 | 0 | 0
  Day 35 DB - Total Cholesterol > ULN | 7 | 8 |  |
  Day 35 DB - Triglycerides > ULN: number analyzed (Participants) | 81 | 78 | 0 | 0
  Day 35 DB - Triglycerides > ULN | 18 | 25 |  |
  End of study - Glucose > ULN: number analyzed (Participants) | 43 | 40 | 21 | 19
  End of study - Glucose > ULN | 6 | 7 | 1 | 3
  End of study - Total Cholesterol > ULN: number analyzed (Participants) | 43 | 40 | 21 | 19
  End of study - Total Cholesterol > ULN | 5 | 4 | 4 | 1
  End of study - Triglycerides > ULN: number analyzed (Participants) | 43 | 40 | 21 | 19
  End of study - Triglycerides > ULN | 8 | 14 | 2 | 4
  Open-label baseline - Glucose > ULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Glucose > ULN |  |  | 6 | 3
  Open-label baseline - Total Cholesterol > ULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Total Cholesterol > ULN |  |  | 1 | 2
  Open-label baseline - Triglycerides > ULN: number analyzed (Participants) | 0 | 0 | 38 | 28
  Open-label baseline - Triglycerides > ULN |  |  | 9 | 6
  Day 14 OL - Glucose > ULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Glucose > ULN |  |  | 5 | 5
  Day 14 OL - Total Cholesterol > ULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Total Cholesterol > ULN |  |  | 3 | 2
  Day 14 OL - Triglycerides > ULN: number analyzed (Participants) | 0 | 0 | 37 | 23
  Day 14 OL - Triglycerides > ULN |  |  | 8 | 3
  Day 84 OL - Glucose > ULN: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84 OL - Glucose > ULN |  |  | 1 | 2
  Day 84 OL - Total Cholesterol > ULN: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84 OL - Total Cholesterol > ULN |  |  | 2 | 1
  Day 84 OL - Triglycerides > ULN: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84 OL - Triglycerides > ULN |  |  | 2 | 2

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Results
Description: Anytime post-baseline includes all assessments from the first dose of study drug until end of study visit in double-blind/open-label part, including unscheduled assessments. Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At study baseline and up to study completion (up to approximately 18 weeks)
Population: All treated participants with available baseline and at least one post-baseline ECG result in the double blind/open-label periods.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 102 | 98 | 38 | 28
Participants
  Baseline - QTcF > 450 msec | 3 | 0 | 3 | 0
  Baseline - QTcF > 480 msec | 0 | 0 | 0 | 0
  Baseline - QTcF > 500 msec | 0 | 0 | 0 | 0
  Baseline - PR ≥ 250 msec | 0 | 0 | 0 | 0
  Baseline - QRS Interval ≥ 150 msec | 0 | 0 | 0 | 0
  Anytime post baseline - QTcF > 450 msec | 2 | 2 | 1 | 0
  Anytime post baseline - QTcF > 480 msec | 0 | 0 | 1 | 0
  Anytime post baseline - QTcF > 500 msec | 0 | 0 | 0 | 0
  Anytime post baseline - QTcF Increase > 30 msec from study baseline | 17 | 21 | 4 | 6
  Anytime post baseline - QTcF Increase > 60 msec from study baseline | 2 | 0 | 0 | 2
  Anytime post baseline - QTcF Increase > 30 msec from open-label baseline: number analyzed (Participants) | 0 | 0 | 38 | 28
  Anytime post baseline - QTcF Increase > 30 msec from open-label baseline |  |  | 4 | 6
  Anytime post baseline - PR ≥ 250 msec | 0 | 0 | 0 | 0
  Anytime post baseline - QTcF Increase > 60 msec from open-label baseline: number analyzed (Participants) | 0 | 0 | 38 | 28
  Anytime post baseline - QTcF Increase > 60 msec from open-label baseline |  |  | 1 | 0
  Anytime post baseline - QRS Interval ≥ 150 msec | 1 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Suicidal Ideation as Defined by a Columbia-Suicide Severity Rating Scale (C-SSRS) Ideation Score of 1 or Greater
Description: The C-SSRS is a clinician- or self-administered questionnaire assessing suicidal ideation and behavior. It rates ideation severity from 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent). It also records the presence or absence of suicidal behaviors, including actual, interrupted, or aborted attempts, and preparatory acts. The highest level of ideation or most severe behavior reported is used to determine suicide risk; higher ideation scores or any suicidal behavior indicate greater risk. Baseline is the last non-missing assessment before first study drug dose.
Time Frame: From first dose to study completion (up to approximately 18 weeks)
Population: All treated participants in the double blind/open-label periods with baseline and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 101 | 97 | 38 | 27
Participants
  Post-Baseline Suicidal ideation (SI) - Any Suicidal Ideation | 7 | 4 | 1 | 3
  Post-Baseline Suicidal ideation - Wish to be Dead | 5 | 4 | 1 | 3
  Post-Baseline Suicidal ideation - Non-Specific Active Suicidal Thoughts | 6 | 3 | 1 | 1
  Post-Baseline SI - Active Suicidal Ideation with any Methods without Intent to Act | 1 | 2 | 0 | 1
  Post-Baseline SI - Active Suicidal Ideation with Some Intent to Act without Specific Plan | 1 | 1 | 0 | 1
  Post-Baseline Suicidal ideation - Active Suicidal Ideation with Specific Plan and Intent | 1 | 0 | 0 | 1

19. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Simpson-Angus Scale (SAS), Barnes Akathisia Rating Scale (BARS), and Abnormal Involuntary Movement Scale (AIMS) Results
Description: Treatment-emergent parkinsonism is defined as Simpson-Angus Scale total score >3 with a baseline score ≤3. Treatment-emergent akathisia is defined as Barnes Akathisia Rating Scale global clinical assessment score >2 with a baseline score ≤2. Treatment-emergent dyskinesia is defined as any Abnormal Involuntary Movement Scale (AIMS) item 1-7 score ≥3 with a baseline score <3 for the item, or score ≥2 on two or more of AIMS items 1-7 with baseline <2 for the items. Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At study baseline, open-label baseline, and up to study completion (up to approximately 18 weeks)
Population: All treated participants in the double blind/open-label periods with baseline and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 102 | 98 | 38 | 28
Participants
  Treatment-Emergent Parkinsonism with respect to study baseline | 3 | 2 | 1 | 1
  Treatment-Emergent Akathisia with respect to study baseline | 2 | 3 | 0 | 0
  Treatment-Emergent Dyskinesia with respect to study baseline | 0 | 2 | 0 | 1
  Treatment-Emergent Parkinsonism with respect to open-label baseline: number analyzed (Participants) | 0 | 0 | 38 | 28
  Treatment-Emergent Parkinsonism with respect to open-label baseline |  |  | 2 | 0
  Treatment-Emergent Akathisia with respect to open-label baseline: number analyzed (Participants) | 0 | 0 | 38 | 28
  Treatment-Emergent Akathisia with respect to open-label baseline |  |  | 0 | 0
  Treatment-Emergent Dyskinesia with respects to open-label baseline: number analyzed (Participants) | 0 | 0 | 38 | 28
  Treatment-Emergent Dyskinesia with respects to open-label baseline |  |  | 0 | 1

20. Secondary Outcome: Change From Baseline in Body Weight
Description: Study baseline is defined as last non-missing assessment prior to the first dose of study drug. Open-label baseline is defined as last non-missing assessment prior to the first dose of study drug in the open-label part.
Time Frame: At study baseline, Day 35 DB, open-label baseline, Day 84 OL, and end of study visit (up to approximately 18 weeks)
Population: All treated participants in the double blind/open-label periods with baseline and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 80 | 80 | 21 | 19
Kg
  Day 35 change from study baseline: number analyzed (Participants) | 80 | 80 | 0 | 0
  Day 35 change from study baseline | -2.125 (2.9596) | -1.184 (3.1079) |  |
  Day 84 change from study baseline: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84 change from study baseline |  |  | -2.889 (6.7846) | -6.955 (5.0021)
  Day 84 change from open-label baseline: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84 change from open-label baseline |  |  | -1.222 (5.2847) | -4.182 (2.9634)
  End of study change from study baseline: number analyzed (Participants) | 44 | 41 | 21 | 19
  End of study change from study baseline | -2.773 (3.1119) | -0.646 (3.3921) | -2.533 (6.4198) | -4.995 (5.2225)
  End of study change from open-label baseline: number analyzed (Participants) | 0 | 0 | 21 | 19
  End of study change from open-label baseline |  |  | -1.462 (5.1589) | -2.850 (3.2432)

21. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: as for outcome 20
Time Frame: At study baseline, Day 35 DB, open-label baseline, Day 84 OL, and end of study visit (up to approximately 18 weeks)
Population: All treated participants in the double blind/open-label periods with baseline and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 80 | 79 | 21 | 19
Kg/m2
  Day 35/Week 5 Change from Study baseline: number analyzed (Participants) | 80 | 79 | 0 | 0
  Day 35/Week 5 Change from Study baseline | -0.79 (1.106) | -0.43 (1.135) |  |
  Day 84/Week 12 Change from Study baseline: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84/Week 12 Change from Study baseline |  |  | -1.10 (2.692) | -2.61 (1.983)
  Day 84/Week 12 Change from open-label baseline: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84/Week 12 Change from open-label baseline |  |  | -0.46 (2.121) | 1.59 (1.276)
  End of Study Change from Study baseline: number analyzed (Participants) | 44 | 41 | 21 | 19
  End of Study Change from Study baseline | -1.01 (1.133) | -0.22 (1.193) | -0.92 (2.499) | -1.83 (1.930)
  End of Study Change from open-label baseline: number analyzed (Participants) | 0 | 0 | 21 | 19
  End of Study Change from open-label baseline |  |  | -0.52 (2.046) | -1.05 (1.224)

22. Secondary Outcome: Change From Baseline in Waist Circumference
Description: as for outcome 20
Time Frame: At study baseline, Day 35 DB, open-label baseline, Day 84 OL, and end of study visit (up to approximately 18 months)
Population: All treated participants in the double blind/open-label periods with baseline and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
Number analyzed (Participants) | 80 | 80 | 21 | 19
cm
  Day 35/Week 5 Change from Study baseline: number analyzed (Participants) | 80 | 80 | 0 | 0
  Day 35/Week 5 Change from Study baseline | -2.27 (4.070) | -1.01 (3.269) |  |
  Day 84/Week 12 Change from Study baseline: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84/Week 12 Change from Study baseline |  |  | -3.96 (8.288) | -4.82 (6.416)
  Day 84/Week 12 Change from open-label baseline: number analyzed (Participants) | 0 | 0 | 18 | 11
  Day 84/Week 12 Change from open-label baseline |  |  | -1.88 (7.198) | -2.27 (4.671)
  End of Study Change from Study baseline: number analyzed (Participants) | 44 | 41 | 21 | 19
  End of Study Change from Study baseline | -3.40 (4.155) | -1.34 (4.167) | -4.69 (8.183) | -3.39 (5.345)
  End of Study Change from open-label baseline: number analyzed (Participants) | 0 | 0 | 21 | 19
  End of Study Change from open-label baseline |  |  | -3.12 (6.874) | -2.45 (2.543)

23. Secondary Outcome: Area Under the Concentration-Time Curve (AUC0-12) of Xanomeline and Trospium - Double-Blind Period
Description: AUC₀-12 (Area Under the Concentration-Time Curve from time zero to 12 hours) is the total amount of drug in the blood measured from the time the drug is given (time zero) up to 12 hours after dosing.
Time Frame: On Day 28 of the Double-Blind Period
Population: All treated participants who received at least one dose of study medicine in the double-blind period and who have available PK data. Prespecified to be reported for the Double-Blind Period only. participants who received treatment are not mutually exclusive
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 42 | 0
pg*h/mL
  Day 28 - Xanomeline 100/20: number analyzed (Participants) | 25 | 0
  Day 28 - Xanomeline 100/20 | 93200 (89.9) |
  Day 28 - Xanomeline 125/30: number analyzed (Participants) | 40 | 0
  Day 28 - Xanomeline 125/30 | 87100 (75.9) |
  Day 28 - Trospium 100/20: number analyzed (Participants) | 28 | 0
  Day 28 - Trospium 100/20 | 48600 (70.4) |
  Day 28 - Trospium 125/30 | 47900 (81.9) |

24. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Xanomeline and Trospium - Double-Blind Period
Description: Cmax is the highest concentration of a drug measured in the blood after it is given.
Time Frame: On Day 28 of the Double-Blind Period
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 45 | 0
pg/mL
  Day 28 - Xanomeline 100/20: number analyzed (Participants) | 28 | 0
  Day 28 - Xanomeline 100/20 | 16000 (129.1) |
  Day 28 - Xanomeline 125/30 | 15900 (95.9) |
  Day 28 - Trospium 100/20: number analyzed (Participants) | 28 | 0
  Day 28 - Trospium 100/20 | 11100 (139.7) |
  Day 28 - Trospium 125/30 | 9330 (99.3) |

25. Secondary Outcome: Time to Cmax (Tmax) of Xanomeline and Trospium - Double-Blind Period
Description: Tmax is the amount of time it takes to reach that highest concentration (Cmax) after the drug is given.
Time Frame: On Day 28 of the Double-Blind Period
Population: as for outcome 23
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo
Number analyzed (Participants) | 45 | 0
Hours
  Day 28 - Xanomeline 100/20: number analyzed (Participants) | 28 | 0
  Day 28 - Xanomeline 100/20 | 1.70 [0.00 to 11.97] |
  Day 28 - Xanomeline 125/30 | 1.93 [0.00 to 11.95] |
  Day 28 - Trospium 100/20: number analyzed (Participants) | 28 | 0
  Day 28 - Trospium 100/20 | 0.56 [0.00 to 11.90] |
  Day 28 - Trospium 125/30 | 0.97 [0.42 to 2.07] |

ADVERSE EVENTS:
Time Frame: Double-blind part: From the start of study drug administration up to week 5. Open-label extension part: From the start of study drug administration up to week 12
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Double-Blind Part: KarXT | Double-Blind Part: Placebo | Open-Label Part: KarXT/KarXT | Open-Label Part: Placebo/KarXT
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/99 | 0/38 | 1/28
Serious Adverse Events (participants affected / at risk) | 0/102 | 3/98 | 0/38 | 3/28
Other Adverse Events (participants affected / at risk) | 97/102 | 90/98 | 33/38 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Part: KarXT (N=102) | Double-Blind Part: Placebo (N=98) | Open-Label Part: KarXT/KarXT (N=38) | Open-Label Part: Placebo/KarXT (N=28)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 2 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Part: KarXT (N=102) | Double-Blind Part: Placebo (N=98) | Open-Label Part: KarXT/KarXT (N=38) | Open-Label Part: Placebo/KarXT (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 2
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 8 | 11 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 4 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 17 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 20 | 2 | 2 | 3
Hyperprolactinaemia (Endocrine disorders) | 4 | 9 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 32 | 20 | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 12 | 3 | 2 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 0 | 2
Nausea (Gastrointestinal disorders) | 38 | 5 | 5 | 14
Retching (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 48 | 2 | 10 | 20
Nasopharyngitis (Infections and infestations) | 5 | 8 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 3 | 2
Alanine aminotransferase increased (Investigations) | 9 | 4 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 6 | 0 | 0
Blood pressure increased (Investigations) | 13 | 4 | 2 | 2
Blood pressure orthostatic decreased (Investigations) | 13 | 9 | 2 | 2
Blood prolactin increased (Investigations) | 4 | 7 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 7 | 5 | 1 | 2
Heart rate increased (Investigations) | 6 | 2 | 1 | 4
Protein urine present (Investigations) | 2 | 1 | 3 | 0
Weight decreased (Investigations) | 21 | 16 | 11 | 10
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4 | 1 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 5 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 8 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 1
Dizziness (Nervous system disorders) | 20 | 5 | 1 | 3
Headache (Nervous system disorders) | 9 | 2 | 0 | 1
Impulsive behaviour (Psychiatric disorders) | 1 | 8 | 2 | 2
Insomnia (Psychiatric disorders) | 6 | 5 | 1 | 2
Schizophrenia (Psychiatric disorders) | 9 | 11 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Hypertension (Vascular disorders) | 8 | 2 | 0 | 3
Orthostatic hypotension (Vascular disorders) | 16 | 14 | 4 | 3
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT05919823/Prot_SAP_000.pdf